CLINICAL TRIAL: NCT06122389
Title: A Double-blinded, Randomized, Multi-center Phase III Clinical Study of SHR2554 Versus Chidamide in Patients With Relapsed/Refractory PTCL
Brief Title: SHR2554 Clinical Study of Chidamide in the Treatment of T-cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR2554-301
Record Dates: First submitted 2023-11-05; First posted 2023-11-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory PTCLT With at Least One Line of Prior Systemic Therapy
MeSH Terms: conditions — Recurrence | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Intervention Model Description: SHR2554 control Chidamide was randomly assigned to either the test group or the control group in a 1:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR2554; Chidamide analog tablets
- Treatment group B (Experimental)
  Interventions: Drug: SHR2554 analog tablets; Chidamide

INTERVENTIONS:
Drug: SHR2554; Chidamide analog tablets — SHR2554 + Chidamide analog tablets
  Arms: Treatment group A
Drug: SHR2554 analog tablets; Chidamide — SHR2554 analog tablets + Chidamide
  Arms: Treatment group B

SUMMARY:
This study was designed to compare the efficacy and safety of SHR2554 with Chidamide in patients with relapsed/refractory PTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old (including 18 and 70 years old), gender is not limited;
2. Histologically confirmed T-cell lymphoma;
3. ECOG physical status must be 0 or 1;
4. Life expectancy ≥12 weeks;
5. For relapsed refractory patients who have received ≥ first-line treatment, at least one prior treatment is adequate;
6. Have not received histone deacetylase inhibitors;
7. Have measurable lesions;
8. Bone marrow function is basically normal;
9. Liver and kidney function is basically normal;
10. Blood coagulation function is basically normal;
11. Female subjects with a possibility of becoming pregnant must undergo a blood pregnancy test prior to the first dose, with a negative result, and be willing to use a highly effective method of contraception for 90 days after signing the notification until the last dose of the study drug. Male subjects whose partners are women at risk of becoming pregnant should be surgically sterilized or agree to use highly effective methods of contraception for 90 days from the date of signing the notification until the last administration of the study drug;
12. The subject has recovered from the toxic effects of the last treatment before the first dosing;
13. The subject personally signs and dates the informed consent to show that the subject has been fully informed of all the circumstances related to the clinical trial;
14. Subjects are willing and able to comply with visit schedules, dosing schedules, laboratory examinations, and other clinical trial procedures.

Exclusion Criteria:

1. Have been treated with compounds with the same mechanism;
2. Accompanied by central nervous system infiltration;
3. Received autologous stem cell transplantation within 60 days before signing the agreement, and received allogeneic stem cell transplantation within 90 days;
4. Major surgery or severe trauma occurred 4 weeks before the first dose of study drug administration;
5. Received anti-tumor treatment within 4 weeks before the first dose of the study drug, and received Chinese medicine treatment with anti-tumor effect within 2 weeks before the first dose of the study drug; Receiving steroid hormones within 7 days prior to the first dose of study drug administration;
6. Active phase of HBV or HCV infection;
7. A history of immunodeficiency, including HIV seropositive, or other acquired or congenital immunodeficiency diseases;
8. Active infection or unexplained fever > 38.5°C within 2 weeks of initial dosing;
9. A history of clinically severe cardiovascular disease;
10. Abnormal electrocardiogram (ECG) examination;
11. Cerebrovascular accident or transient ischemic attack occurred within 6 months before entering the study;
12. Have other malignancies within 5 years prior to screening, other than adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery (allowing hormone therapy for non-metastatic prostate cancer or breast cancer), and papillary thyroid cancer;
13. The subject has another serious/severe acute or chronic illness or mental illness, including recent (within the past year) or current suicidal ideation or behavior, or laboratory abnormalities that may increase the risks associated with participation in the study or administration of the investigational drug, may interfere with the interpretation of the study results, or may interfere with the investigator's judgment;
14. The subjects are the staff of the research center directly related to this clinical trial or their family members, or the subordinates of this trial although not directly related to this trial, or the staff employed by the sponsor directly related to this trial;
15. Pregnant and lactating women;
16. The subject is unable to swallow, or has a history of active gastrointestinal inflammation, chronic diarrhea, known diverticulosis, or a history of gastrectomy or gastric banding that affects drug absorption;
17. The subject is taking a known medium or strong CYP inducer;
18. In the judgment of the investigator, objective conditions (including the subject's psychological state, family relationship, social factors or geographical factors) make the subject unable to complete the planned study or the subject has other factors, concomitant diseases, combined treatment or abnormal laboratory examination that may lead to the forced termination of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by IRC | up to 3 years

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided